CLINICAL TRIAL: NCT00604292
Title: Evaluation of the PillCam Colon Capsule Endoscopy Preparation and Procedure
Brief Title: Evaluation of the PillCam Colon Capsule Endoscopy (PCCE) Preparation and Procedure
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: MA-102
Record Dates: First submitted 2008-01-29; First posted 2008-01-30 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2010-03

CONDITIONS: Colonic Diseases
Keywords: Colonic Diseases
MeSH Terms: conditions — Colonic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Patients that are indicated for colonoscopy, who are suspected or known to suffer from colonic diseases

SUMMARY:
To evaluate the effect of a modified preparation and procedure on colon cleansing level

DETAILED DESCRIPTION:
The evaluation of subjects with suspected colonic disease includes endoscopic imaging by colonoscopy and radiologic imaging such as air-contrast barium enema, abdominal/pelvic CT, or virtual colonoscopy. The Given® Diagnostic System offers an alternative approach for endoscopic visualization of the colon using capsule endoscopy, a swallowable device which contains imagers, light sources, a power source and a RF transmitter. Advantages of the Given® Diagnostic System include the elimination of the need for conscious sedation, the minimally invasive, painless nature of the exam, and the ability to pursue normal daily activities immediately following the procedure . Furthermore, compared to standard colonoscopy, the Given® Diagnostic System may be more readily accepted by the subjects, thereby improving subjects' willingness to undergo a diagnostic evaluation of the colon and comply with colorectal cancer screening recommendations.

The PillCam™ SB capsule (formerly M2A® Capsule) that was FDA-approved in August 2001 for small bowel evaluation has been ingested to date by more than 300,000 people worldwide and is well accepted by patients and physicians as well as the processional societies. However, adequate visualization of the colon cannot be achieved with the standard PillCam™ SB capsule because of the anatomical and physiological properties of the colon which are significantly different than the small bowel. Moreover, other issues that limit the evaluation of the colonic mucosa by the standard PillCam™ SB procedure include an unsatisfactory level of colon cleanliness and slow progression of the PillCam™ SB capsule through the colon during the desired examination time. Therefore, the development and introduction of a specially designed, customized colon capsule combined with a dedicated capsule colonoscopy procedure protocol will allow for more efficient evaluation of the colonic mucosa. This is expected to improve the capability of the Given® Diagnostic System to detect colonic pathologies and to serve as a diagnostic and screening tool for colonic disease. Further details of the PillCam™ Colon Capsule Endoscope (PCCE) can be found in the device description section.

This is a pilot study that is designed to compare capsule colonoscopy and colonoscopy procedures with respect to colon cleansing level and progression of colon capsule. Furthermore, the two procedures will be compared in regards to the detection of colon abnormalities.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study:

* Subject is between the ages of 18-75 years.
* Subject is suspected/known to suffer from large bowel disease and was clinically referred for colonoscopy (rectal bleeding, melena, positive FOBT, recent change of bowel habits, CRC screening, UC, positive findings on a GI radiographic study)

Exclusion Criteria:

The presence of any of the following will exclude a subject from study enrollment:

* Subject has dysphagia or any swallowing disorder
* Subject has Congestive heart failure
* Subject is known to suffer from diabetes
* Subject has high degree of renal insufficiency
* Subject has had prior abdominal surgery of the gastrointestinal tract other than uncomplicated procedures that would be unlikely to lead to bowel obstruction based on the clinical judgment of the investigator
* Subject has a cardiac pacemakers or other implanted electromedical devices.
* Subject has any allergy or other known contraindication to the medications used in the study
* Subject is expected to undergo MRI examination within 7 days after ingestion of the capsule.
* Subject with high risk for capsule retention: Crohn's disease, SB tumors, radiation enteritis, NSAID, surgical anastomosis,
* Subject has any condition, which precludes compliance with study and/or device instructions.
* Women who are either pregnant or nursing at the time of screening, who intend to be during the study period, or are of child bearing potential and do not practice medically acceptable methods of contraception
* Subject suffers from life threatening conditions
* Subject currently participating in another clinical study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that are indicated for colonoscopy, who are suspected or known to suffer from colonic diseases
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2007-06; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Colon cleansing level score | within 7 days

SECONDARY OUTCOMES:
Accuracy parameters of PCCE, compared to colonoscopy | within 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Riemann, Prof. Dr., Principal Investigator — Klinikum Ludwigshafen gGmbH
Locations (3):
- Germany (3):
  - Klinikum Ludwigshafen gGMBH, Ludwigshafen, Bremserster 79
  - Evangelisches Krankenhaus, Düsseldorf
  - Allgemeines Krankenhaus Altona, Hamburg